CLINICAL TRIAL: NCT03677544
Title: Predictive Factorsfor Final Pathologic Ureteral Sections on 700 Radical Cystectomy Specimens: Implicationsforintraoperativefrozensection Decision-making
Brief Title: Predictive Factorsfor Final Pathologic Ureteral Sections
Acronym: CYSTECTOMEN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0051
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2018-09

CONDITIONS: Urothelial Carcinoma
Keywords: radical systectomy; Ureteral frozen section
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- no intraoperative FS examination: Surgery was performed through either open or laparoscopic approach with an extended pelvic lymph node dissection up to the common iliac bifurcation. procedures were performed between 1980 and 2013
  Interventions: Other: laparoscopic approach with an extended pelvic lymph
- intraoperative FS examination: Surgery was performed through either open or laparoscopic approach with an extended pelvic lymph node dissection up to the common iliac bifurcation procedures were performed between 2001 and 2013
  Interventions: Other: laparoscopic approach with an extended pelvic lymph

INTERVENTIONS:
Other: laparoscopic approach with an extended pelvic lymph — Surgery was performed through either open or laparoscopic approach with an extended pelvic lymph node dissection up to the common iliac bifurcation

SUMMARY:
To identify preoperative predictive factors for final ureteral section invasion after radical cystotomie (RC) and to validate significant factors on an external independent cohort. The investigators retrospectively reviewed data of all consecutive RC performed for bladder cancer in 2 high-volume institutions. Clinical, pathological, and follow-up data were collected prospectively and reviewed retrospectively. Pathological evaluation was performed by 2 well-trained uropathologists in each center. Logistic regression analyses were performed to identify predictive factors for final ureteral sections involvement. Significant factors in cohort A were validated in cohort B. Receiver operating curve and area under curve were modeled to evaluate predictive accuracy of the markers

DETAILED DESCRIPTION:
To identify preoperative predictive factors for final ureteral section invasion after radical cystotomie (RC) and to validate significant factors on an external independent cohort. Pathological evaluation was performed by 2 well-trained uropathologists in each center (Y.A. and C.C). The investigators retrospectively reviewed data of all consecutive RC performed for bladder cancer in 2 high-volume institutions. Clinical, pathological, and follow-up data were collected prospectively and reviewed retrospectively. Pathological evaluation was performed by 2 well-trained uropathologists in each center. Logistic regression analyses were performed to identify predictive factors for final ureteral sections involvement. Significant factors in cohort A were validated in cohort B. Receiver operating curve and area under curve were modeled to evaluate predictive accuracy of the markers

ELIGIBILITY:
Inclusion Criteria:

* patients > 18 years
* patients reoperative predictive factors for final ureteral section invasion after radical cystectomy

Exclusion Criteria:

* patients < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In cohort A, most patients did not have intraoperative FS examination although it was performed in some cases depending on the surgeon's habits (N¼92). All patients had intraoperative FS in the validation cohort B. All cystectomies performed for nononcological purposes were excluded. All patients had nonmetastatic bladder cancer on preoperative computed tomography (CT) scans.
Sampling Method: Non-Probability Sample
Enrollment: 748 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
preoperative predictive factors | 2years
  The objective of this study is to identify preoperative predictive factors for final ureteral section invasion after radical cystectomy (RC) and to validate significant factors on an external independent cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Saint, MD, PhD, Principal Investigator — CHU AMIENS

IPD SHARING:
Plan to Share IPD: No